CLINICAL TRIAL: NCT06209684
Title: Carbofix Pedicle Screw System: Randomized Clinical Trial to Evaluate the Clinical and Radiographic Outcomes of the Use of a Carbon Fiber Device Compared to Titanium Devices in Patients Undergoing Spinal Arthrodesis for Degenerative Spinal Diseases
Brief Title: Carbofix Pedicle Screw System: Evaluation of the Clinical and Radiographic Outcomes of the Use of a Carbon Fiber Device Compared to Titanium Devices in Patients Undergoing Spinal Arthrodesis for Degenerative Spinal Diseases
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Istituto Ortopedico Rizzoli (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Carbofix degenerative
Record Dates: First submitted 2024-01-04; First posted 2024-01-17 (Actual); Last update posted 2025-01-17 (Actual); Status verified 2025-01

CONDITIONS: Degenerative Disc Disease
Keywords: degenerative spine disease
MeSH Terms: conditions — Intervertebral Disc Degeneration | interventions — Titanium

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental (Experimental): CarboFix implant for spinal surgery
  Interventions: Procedure: Carbofix
- Traditional (Active Comparator): Titanium implant for spinal surgery
  Interventions: Procedure: Titanium

INTERVENTIONS:
Procedure: Titanium — Spinal stabilization using titanium screws and rods
  Arms: Traditional
Procedure: Carbofix — Spinal stabilization using CarboFix screws and rods
  Arms: Experimental

SUMMARY:
Previous clinical study carried out on cancer patients at IOR Spine Surgery (approved in October 2014). The carbon device is indicated in patients suffering from vertebral tumors who need stabilization and will then carry out radiotherapy, because carbon has a practically zero level of interference with ionizing radiation. Carbon also allows for better visualization of the implants on MRI/CT and X-ray. There are no studies in the literature analyzing the use of carbon fiber devices in lumbar degenerative pathologies.

118 patients suffering from degenerative spinal pathology requiring 1 or 2 levels of lumbar or lumbosacral fusion will be valutated.

ELIGIBILITY:
Inclusion Criteria:

* Patients suffering from degenerative spinal pathology or spondylolisthesis who require instrumented stabilization on 1-2 levels;
* Age greater than or equal to 18 years;
* Ability to understand and sign the informed consent to the study and to follow the required follow-ups.

Exclusion Criteria:

* Metabolic bone disease.
* History of Paget's disease or other osteodystrophies, whether acquired or congenital, including renal osteodystrophy, hyperthyroidism, hypothyroidism, Ehlers-Danlos syndrome, osteogenesis imperfecta, achondroplasia.
* Neoplastic disease.
* History of mental disorder or current psychiatric treatment.
* Pregnancy.
* Immunodeficiency diseases.
* Infectious bone disease (discitis, osteomyelitis)
* Treatment with drugs that can interfere with bone metabolism
* Inability to understand and sign the informed consent to the study and to follow the required follow-up visits.
* Alcohol and/or drug abuse
* Obesity
* Metal allergy
* Participation in other studies on drugs or devices (within 30 days)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 118 (Estimated)
Dates: Start 2022-04-29 (Actual); Primary Completion 2026-04-29 (Estimated); Study Completion 2027-04-29 (Estimated)

PRIMARY OUTCOMES:
Fusion rate | through study completion, an average of 1 year
  Fusion rate after 12 months as demonstrated by computed tomography scan (CT scan).
  The CT scan will be evaluated by Brantigan scale.

SECONDARY OUTCOMES:
Classification system of surgical complications specific for spine | at baseline (day 0)
  rate of intra-operative complications evaluated by SAVES classification system specific for spine
Classification system of surgical complications specific for spine | up to 12 months
  rate of post-operative complications evaluated by SAVES classification system specific for spine
Visual Analogue Scale | at baseline (day 0)
  A Visual Analogue Scale (VAS) is one of the pain rating scales used for the first time in 1921 by Hayes and Patterson. It is often used in epidemiologic and clinical research to measure the intensity or frequency of various symptoms.
Visual Analogue Scale | after 12 months
  A Visual Analogue Scale (VAS) is one of the pain rating scales used for the first time in 1921 by Hayes and Patterson. It is often used in epidemiologic and clinical research to measure the intensity or frequency of various symptoms.
Visual Analogue Scale | after 3 months
  A Visual Analogue Scale (VAS) is one of the pain rating scales used for the first time in 1921 by Hayes and Patterson. It is often used in epidemiologic and clinical research to measure the intensity or frequency of various symptoms.
Visual Analogue Scale | after 6 months
  A Visual Analogue Scale (VAS) is one of the pain rating scales used for the first time in 1921 by Hayes and Patterson. It is often used in epidemiologic and clinical research to measure the intensity or frequency of various symptoms.
Oswestry Disability Index | at baseline (day 0)
  The Oswestry Disability Index (ODI) is a self-administered and validated questionnaire in Italian which aims to evaluate disabilities in subjects suffering from low back pain in both the acute and chronic phases.
Oswestry Disability Index | after 12 months
  The Oswestry Disability Index (ODI) is a self-administered and validated questionnaire in Italian which aims to evaluate disabilities in subjects suffering from low back pain in both the acute and chronic phases.
Oswestry Disability Index | after 3 months
  The Oswestry Disability Index (ODI) is a self-administered and validated questionnaire in Italian which aims to evaluate disabilities in subjects suffering from low back pain in both the acute and chronic phases.
Oswestry Disability Index | after 6 months
  The Oswestry Disability Index (ODI) is a self-administered and validated questionnaire in Italian which aims to evaluate disabilities in subjects suffering from low back pain in both the acute and chronic phases.
EuroQoL-5D | at baseline (day 0)
  EQ-5D is a standardised measure of health-related quality of life developed by the EuroQol Group to provide a simple, generic questionnaire for use in clinical and economic appraisal and population health surveys. EQ-5D assesses health status in terms of five dimensions of health and is considered a 'generic' questionnaire because these dimensions are not specific to any one patient group or health condition
EuroQoL-5D | after 12 months
  EQ-5D is a standardised measure of health-related quality of life developed by the EuroQol Group to provide a simple, generic questionnaire for use in clinical and economic appraisal and population health surveys. EQ-5D assesses health status in terms of five dimensions of health and is considered a 'generic' questionnaire because these dimensions are not specific to any one patient group or health condition
EuroQoL-5D | after 3 months
  EQ-5D is a standardised measure of health-related quality of life developed by the EuroQol Group to provide a simple, generic questionnaire for use in clinical and economic appraisal and population health surveys. EQ-5D assesses health status in terms of five dimensions of health and is considered a 'generic' questionnaire because these dimensions are not specific to any one patient group or health condition
EuroQoL-5D | after 6 months
  EQ-5D is a standardised measure of health-related quality of life developed by the EuroQol Group to provide a simple, generic questionnaire for use in clinical and economic appraisal and population health surveys. EQ-5D assesses health status in terms of five dimensions of health and is considered a 'generic' questionnaire because these dimensions are not specific to any one patient group or health condition
Short Form-12 | at baseline (day 0)
  The SF-12 is composed of 12 items (derived from the 36 of the original SF-36 questionnaire) which produce two measures relating to two different aspects of health: physical health and mental health.
  The SF-12 is made up of 4 scales (physical functioning, role and physical health, role and emotional state, mental health) measured by 2 items each and 4 scales each measured by one item (physical pain, vitality, social activities and general health).
Short Form-12 | after 12 months
  The SF-12 is composed of 12 items (derived from the 36 of the original SF-36 questionnaire) which produce two measures relating to two different aspects of health: physical health and mental health.
  The SF-12 is made up of 4 scales (physical functioning, role and physical health, role and emotional state, mental health) measured by 2 items each and 4 scales each measured by one item (physical pain, vitality, social activities and general health).
Short Form-12 | after 3 months
  The SF-12 is composed of 12 items (derived from the 36 of the original SF-36 questionnaire) which produce two measures relating to two different aspects of health: physical health and mental health.
  The SF-12 is made up of 4 scales (physical functioning, role and physical health, role and emotional state, mental health) measured by 2 items each and 4 scales each measured by one item (physical pain, vitality, social activities and general health).
Short Form-12 | after 6 months
  The SF-12 is composed of 12 items (derived from the 36 of the original SF-36 questionnaire) which produce two measures relating to two different aspects of health: physical health and mental health.
  The SF-12 is made up of 4 scales (physical functioning, role and physical health, role and emotional state, mental health) measured by 2 items each and 4 scales each measured by one item (physical pain, vitality, social activities and general health).

CONTACTS AND LOCATIONS:
Locations (1):
- Istituto Ortopedico Rizzoli, Bologna, Italy

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- [Background] Boriani S, Tedesco G, Ming L, Ghermandi R, Amichetti M, Fossati P, Krengli M, Mavilla L, Gasbarrini A. Carbon-fiber-reinforced PEEK fixation system in the treatment of spine tumors: a preliminary report. Eur Spine J. 2018 Apr;27(4):874-881. doi: 10.1007/s00586-017-5258-5. Epub 2017 Aug 16. PMID 28815357
- [Background] Boriani S, Pipola V, Cecchinato R, Ghermandi R, Tedesco G, Fiore MR, Dionisi F, Gasbarrini A. Composite PEEK/carbon fiber rods in the treatment for bone tumors of the cervical spine: a case series. Eur Spine J. 2020 Dec;29(12):3229-3236. doi: 10.1007/s00586-020-06534-0. Epub 2020 Jul 20. PMID 32691220
- [Result] Vaccaro AR, Garfin SR. Pedicle-Screw Fixation in the Lumbar Spine. J Am Acad Orthop Surg. 1995 Oct;3(5):263-274. doi: 10.5435/00124635-199509000-00002. PMID 10795032